CLINICAL TRIAL: NCT00002920
Title: A Randomized Comparison Of Medroxyprogesterone Acetate (MA) And Observation For Prevention Of Endometrial Pathology In Postmenopausal Breast Cancer Patients Treated With Tamoxifen, Phase III
Brief Title: S9630, Medroxyprogesterone in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000065314; CALGB-49901 (Other: CALGB); S9630 (Other: SWOG); U10CA037429 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Breast Cancer; Endometrial Cancer
Keywords: endometrial cancer; stage I breast cancer; stage II breast cancer; ductal breast carcinoma in situ; lobular breast carcinoma in situ; Paget disease of the breast
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Paget's Disease, Mammary | interventions — Medroxyprogesterone; Tamoxifen; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tamoxifen alone (Active Comparator): Tamoxifen alone x 5 years
  Interventions: Drug: tamoxifen citrate; Procedure: adjuvant therapy
- Tamoxifen plus MPA (Experimental): Tamoxifen Plus Medroxyprogesterone Acetate (MPA) x 5 years
  Interventions: Drug: medroxyprogesterone; Drug: tamoxifen citrate; Procedure: adjuvant therapy

INTERVENTIONS:
Drug: medroxyprogesterone
  Arms: Tamoxifen plus MPA
Drug: tamoxifen citrate
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: It is not yet known whether medroxyprogesterone is effective in preventing endometrial disorder in patients with breast cancer who are taking tamoxifen.

PURPOSE: Randomized phase III trial to study the effectiveness of medroxyprogesterone in preventing endometrial disorder in postmenopausal women who have ductal carcinoma in situ, lobular carcinoma in situ, Paget's disease of the nipple, stage I breast cancer, or stage II breast cancer and who are taking tamoxifen.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare endometrial pathologic diagnoses (proliferative changes, simple or cystic hyperplasia, complex adenomatous hyperplasia, hyperplasia with atypia, and carcinoma) in postmenopausal women with breast carcinoma treated with adjuvant tamoxifen who are randomly assigned to medroxyprogesterone acetate (MA) vs observation.
* Compare endometrial pathologic diagnoses (persistent endometrial hyperplasia, atypia, or carcinoma) resulting in tamoxifen discontinuation and intermittent bleeding in patients treated with these regimens.
* Characterize the incidence of spontaneous regression and progression of simple or cystic hyperplasia in these patients.
* Characterize endometrial biopsy results using different endometrial stripe width cut-off points, for cases in which the width is at least 5 mm by endovaginal ultrasound in patients receiving tamoxifen.
* Compare changes over time in endometrial oncogene expression (e.g., c-fos, c-jun, p53, IGF1) and receptor status in patients receiving tamoxifen with or without prior chemotherapy who are randomly assigned to MA vs observation.
* Describe the associations among change in gene expression, receptor status, endometrial abnormality, length of tamoxifen exposure, and prior chemotherapy in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to adjuvant chemotherapy (yes vs no), number of positive nodes (0-3 vs at least 4), and endovaginal sonogram endometrial stripe (less than 5 mm vs at least 5 mm). Patients are randomized to 1 of 2 arms.

All patients receive adjuvant oral tamoxifen daily for five years.

* Arm I: Patients undergo observation.
* Arm II: Patients receive oral medroxyprogesterone acetate on days 1-14. Treatment repeats every 3 months for 5 years.

Patients are followed every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 330 patients (165 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following histologically proven diagnoses:

  * Primary invasive adenocarcinoma of the unilateral or bilateral breast

    * Stage I, IIA, or IIB (T1-3, N0-1, M0)
    * No recurrent invasive breast cancer
  * Ductal carcinoma in situ (DCIS)
  * Lobular carcinoma in situ (LCIS) with microinvasion
  * Paget's disease of the nipple
* No sarcoma, lymphoma, or apocrine, adenocystic, or squamous cell cancer of the breast
* Currently free of breast cancer (no evidence of disease)

  * No evidence of distant disease on chest x-ray or chest CT scan and mammogram of the opposite breast within the past year
* Prior definitive local treatment of primary lesion (mastectomy or breast-sparing procedure with radiotherapy) and either axillary node or sentinel node biopsy

  * Surgical margins clear of both infiltrating carcinoma (any type) and DCIS

    * No gross or microscopically positive margins except:

      * Invasive cancer or DCIS at the focal margin treated with definitive radiotherapy
      * Gross or LCIS at the final margin
  * Biopsy requirement waived for DCIS or LCIS with minimal microinvasion
* Patients with breast-sparing procedure must have received or be planning to receive radiotherapy at start of tamoxifen treatment
* No endometrial simple or cystic hyperplasia, proliferative changes, complex (adenomatous) or atypical hyperplasia, or carcinoma
* Patients must be planning one of the following:

  * Starting adjuvant tamoxifen for five years OR
  * Started tamoxifen within 28 days prior to study and planning to receive adjuvant tamoxifen for five years
* Hormone receptor status:

  * Candidate for adjuvant tamoxifen therapy

PATIENT CHARACTERISTICS:

Age:

* Adult

Sex:

* Female

Menopausal status:

* Postmenopausal defined as:

  * At least 1 year since last menstrual period
  * At least 2 months since bilateral oophorectomy prior to breast cancer diagnosis
  * 4-12 months since last menstrual period and FSH elevated to postmenopausal range
  * Postmenopausal estrogen therapy and 55 years of age or older

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Fertile patients must use effective contraception during and for at least 2 months after study
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or stage I or II cancer currently in complete remission
* No concurrent nonmalignant-related illness that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Adjuvant chemotherapy allowed
* No concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* No prior hormonal treatment for breast cancer (except tamoxifen)
* No concurrent postmenopausal estrogen therapy

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics
* No prior or concurrent hysterectomy

Other:

* No prior or current participation in an adjuvant intergroup trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 1997-03; Primary Completion 2006-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Endometrial pathologic diagnosis | 2 years after registration
  Endometrial pathologic diagnosis at 2 years after registration

SECONDARY OUTCOMES:
Endometrial pathologic diagnosis | 5 years after registration
  Endometrial pathologic diagnosis at 5 years after registration

CONTACTS AND LOCATIONS:
Overall Officials: Ronald K. Potkul, MD, Study Chair — Loyola University; Barbara L. Smith, MD, PhD, Study Chair — Massachusetts General Hospital
Locations (122):
- United States (122):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - Loma Linda (Pettis), Loma Linda, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - Naval Medical Center - San Diego, San Diego, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield, Southfield, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - St. Louis University Hospital Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - North Shore University Hospital, Manhasset, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - NorthEast Oncology Associates - Concord, Concord, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital at Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Tennessee Cancer Institute at Methodist Central Hospital, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Incorporated - Roanoke, Roanoke, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington